CLINICAL TRIAL: NCT04608097
Title: Understanding Reactions to Emotional Material in the Media During COVID-19 and the Connections to Cognitive Activities
Brief Title: Understanding Reactions to Emotional Material in the Media During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Emily Holmes, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020-03991
Record Dates: First submitted 2020-10-28; First posted 2020-10-29 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Healthy Participants; Intrusive Memories
Keywords: Digital Intervention; Intrusive Memories; Trauma Film Paradigm; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple cognitive task intervention (Experimental): A memory cue followed by playing the computer game "Tetris" (on own smartphone) with mental rotation instructions for ca. 12 minutes.
  Interventions: Behavioral: Simple cognitive task intervention
- Attention placebo (Placebo Comparator): A memory cue followed by listening to a podcast (on own smartphone) for ca. 12 minutes.
  Interventions: Behavioral: Attention Placebo

INTERVENTIONS:
Behavioral: Simple cognitive task intervention — A memory cue followed by playing the computer game "Tetris" (on own smartphone) with mental rotation instructions for ca. 12 minutes.
  Arms: Simple cognitive task intervention
Behavioral: Attention Placebo — A memory cue followed by listening to a podcast (on own smartphone) for ca. 12 minutes.
  Arms: Attention placebo

SUMMARY:
This feasibility study aims to adapt a protocol usually run in the laboratory in the Psychology Department for healthy participants (including the trauma film paradigm (James et al., 2016) and a simple cognitive task intervention) to remote (online) delivery. The motivation for this was restrictions to running in person laboratory experiments during the COVID-19 pandemic.

Participants will view film footage with COVID-19 related and potentially traumatic content (e.g. of seriously ill or dying patients in hospitals). Following film viewing, participants will be randomly allocated to either the experimental condition (simple cognitive task intervention, i.e. a memory cue followed by playing the computer game "Tetris" with mental rotation instructions) or the control condition (attention placebo, i.e., a memory cue followed by listening to a podcast for a similar duration). Any intrusive memories induced by the film (analogue trauma) will be monitored in a daily diary. It is predicted that the film (analogue trauma) will generate intrusive memories. If intrusive memories are generated, then it is predicted that participants in the experimental condition will report fewer intrusive memories related to the film (analogue trauma) during the following week than participants in the control condition.

The development of this paradigm may inform the future development of a simple technique to prevent intrusive memories e.g. after repeated media consumption related to the COVID-19 pandemic.

DETAILED DESCRIPTION:
This is a between-groups experimental study with healthy participants informed by prior laboratory work. It includes two sessions and a seven-day daily diary in between sessions. In this feasibility study, for the first time all study procedures will be delivered remotely rather than in a laboratory because of the COVID-19 pandemic. The primary outcome is the number of intrusive memories related to the film (analogue trauma) recorded in a daily electronic diary during the following week (week 1).

The first aim is to investigate if the film (analogue trauma) will generate intrusive memories. The second aim is, if intrusive memories are generated, to investigate if participants in the experimental condition will report fewer intrusive memories of the film (analogue trauma) than participants in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Fluent in spoken and written Swedish
* Willing to watch a video containing emotional, distressing footage
* Have access to an internet enabled smartphone/computer

Exclusion Criteria:

* Have participated in a study in which similar stimuli were used
* Currently receiving treatment for a mental health problem (e.g. depression, anxiety, ADHD, addiction), including psychological therapy, counselling or medication
* Neurological illness (e.g., epilepsy)
* Planning to undertake a stress-inducing examination (e.g. university examination or driving test) during the week of study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories related to the trauma film | Week 1
  Number of intrusive memories related to the trauma film recorded by participants in a brief diary daily for 7 days.

SECONDARY OUTCOMES:
Characteristics of intrusive trauma memories related to the trauma film | Week 1
  2 self-rated items measuring the level of distress and vividness associated with the intrusions related to the trauma film (11-point scales from 0 to 10) rated within the diary. High scores indicate higher level of distress/vividness.
Intrusion questionnaire | Week 1 follow-up
  1 self-rated item measuring the frequency of intrusive/unwanted memories of the trauma film in the previous week on a 7-point scale (from "never" to "many times a day", with a follow-up question to specify the number if necessary). Unless the answer to item 1 is "never", 5 self-rated items measuring the characteristics of intrusive/unwanted memories in the previous week. The level of distress, nowness, reliving, disconnectedness and whether different triggers are associated with the intrusive/unwanted memories of the trauma film are measured on a 101-point scale (from 0 to 100). Higher scores indicate more intrusive/unwanted memories, higher levels of distress/nowness/reliving/disconnectedness and a greater number of different triggers.
Impact of Event Scale - Revised (IES-R): Degree of subjective distress of post-film intrusions | Week 1 follow-up
  Self-report measure that assesses subjective distress after a traumatic event (with reference to the trauma film). Here we include the intrusion subscale (8 items). Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Items are summed (subscale score ranges from 0 to 32). Higher scores indicate worse outcome.
Self-rated functioning associated with intrusive memories | Week 1 follow-up
  A single bespoke item on impact on daily functioning associated with the intrusions from the trauma film rated on a 11-point scale (from 0 "none"; 5 "some"; 10 "extreme"). Higher scores indicate higher level of functional impairment.
Self-rated concentration disruption associated with intrusive memories | Week 1 follow-up
  A single bespoke item measuring the level of concentration disruption associated with the intrusions from the trauma film (11 point scale from 0 to 10). High scores indicate higher level of concentration disruption.
Self-rated sleep ratings | Week 1 follow-up
  Two self rated items: Item 1 measures the extent of being troubled by poor sleep (with reference to study event) on a 5-point scale (from not at all to very much), and item 2 measures the number of nights in the week with sleep problems on a 5-point scale (from 0-1 to 5-7 nights). Each 5-point scale is reverse scored (4 - 0) then summed. Possible total scores range from 0 - 8, with higher values indicative of better sleep.
Behavior Change Questionnaire | Week 1 follow-up
  7 bespoke self-report items assessing how much the trauma film affected related safety and avoidance behaviors from 0 (not at all) to 100 (extremely) (e.g. "I took greater care to keep a distance in public places"). A free text response field for other behaviors that were affected by the trauma film.
Intrusion provocation task (IPT) | Week 1 follow-up
  In the Intrusion Provocation Task (IPT), participants are presented with neutral still images from the trauma film. Immediately afterwards for the next two minutes, they are allowed to think freely and report intrusions by pressing a button. The IPT intrusion score is calculated by the total frequency of intrusions (i.e. number of button presses), whilst higher values represent more intrusions.
Verbal recognition memory test | Week 1 follow-up
  The verbal recognition memory test comprises a number of true/false written statements relating to the trauma film. Participants indicate true or false as to whether or not the written statement about the film they watched 7 days earlier is correct. The score is the sum of correct responses, a higher score indicating better verbal recognition memory of the trauma film.
Visual recognition memory test | Week 1 follow-up
  The visual recognition memory test consists of static visual images - some are taken from throughout the film (different images from those used in the IPT), and some are unviewed images presented as filler. Images are presented individually and participants are instructed to view each image for 5 s. Participants indicate yes or no as to whether or not they recognize the image as being from the trauma film they watched 7 days earlier. The score is the sum of correct responses, a higher score indicating better visual recognition memory of the trauma film.
Time perspective questionnaire | Week 1 follow-up
  8 self-report items (5-point scale from 1 to 5) measuring time perspective on three subscales: past perspective (items 3, 5, 7), present perspective (items 1, 8) and future perspective (items 2, 4, 6). Item scores for each subscale will be summed. Higher values indicate higher levels of past/present/future time perspective.
Future self questionnaire | Week 1 follow-up
  Three free text response fields asking to imagine a future self identity in relation to social/occupational/other important situations. A single item measuring which of these future identities has been most affected by the COVID-19 pandemic. Then a free text response field to describe a mental image of this identity, 4 items measuring vividness (1 "not vivid at all", 10 "very vivid"), positivity (1 "very negative", 10 "very positive"), regularity of rehearsal (1 "never", 10 "very regularly"), and likelihood (1 "not at all likely", 10 "very likely") of that image on a 10-point scale. 3 items measuring the perspective of viewing that mental image ("through own eyes" or "as if seeing oneself"), whether other people are in the image (if yes, how many), and how old one will be in the image. All items are answered in terms of how the image was before and after the COVID-19 pandemic. Free text response field asking how the COVID-19 pandemic affected the future identity image.
Future Expectancy Scale | Week 1 follow-up
  Self-report measure that assesses expectancies about positive future life events. 10 items are rated regarding how likely it is that the event will happen in one's future on a 7-point scale ranging from 1 ("not at all likely") to 7 ("extremely likely"). Items are summed. Higher scores indicate more optimistic/positive future expectancies.

OTHER OUTCOMES:
Number of unwanted/intrusive memories of COVID-19 media footage during the week before study participation | Day 1
  1 self-rated item measuring the frequency of intrusive/unwanted memories of traumatic events related to COVID-19 or media consumption on COVID-19 in the previous week on a 7-point scale (from "never" to "many times a day", with a follow-up question to specify the number if necessary).
Negative mood ratings | Day 1 and Week 1 follow-up
  6 visual analogue scale ratings measuring how sad, hopeless, depressed, fearful, horrified and anxious participants feel "right at this very moment" on a scale from 1 "not at all" to 10 "extremely" assessed before and after film viewing and after completing the experimental or control condition task as well as in the beginning of session 2 (Week 1 follow-up). Rating are summed yielding a composite negative mood score, with higher scores indicating higher negative mood.
Post-trauma-film ratings | Day 1
  4 rating scales measuring how distressing participants found the trauma film, how much attention they paid to the film, how personally relevant the film was for them and how much they looked away from the film on a 11-point scale from 0 "not at all" to 10 "extremely".
Hotspots related to the trauma film (memory cue) | Day 1
  6 free text response fields in which participants are asked to list the images/moments of the trauma film that were worst for them with a brief description. This list is part of the memory cue procedure in the experimental/control condition.
Post-condition ratings | Day 1
  4 rating scales measuring how entertaining/difficult/distracting participants found the task they were doing in the experimental/control condition and how much attention they paid to the task they were doing in the experimental/control condition on a 11-point scale from 0 "not at all" to 10 "extremely".
Demand ratings about conditions | Week 1 follow-up
  2 items measuring to which extent participants believe that playing Tetris/listening to a podcast after watching a distressing film increases or decreases intrusive memories of the film on a 21-point scale from -10 (extreme decrease), 0 (no effect), to 10 (extreme increase).
Perceived Awareness of the Research Hypothesis Scale | Week 1 follow-up
  4 items measuring to which extent participants agree to statements about being aware of the purpose of the study on a 7-point scale from 1 "Do not agree at all" to 7 "Completely agree". Two items are reverse scored and then all items are summed. Higher scores indicate higher demand effects.
Exposure to COVID-19 related media in the week of study participation | Week 1 follow-up
  5 items measuring the number of hours (0-11 or more) per day during the previous week that participants consumed COVID-19 related media content on TV, radio, newspaper, online news, or social media.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Holmes, Prof, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

REFERENCES:
- [Result] James EL, Lau-Zhu A, Clark IA, Visser RM, Hagenaars MA, Holmes EA. The trauma film paradigm as an experimental psychopathology model of psychological trauma: intrusive memories and beyond. Clin Psychol Rev. 2016 Jul;47:106-42. doi: 10.1016/j.cpr.2016.04.010. Epub 2016 Apr 21. PMID 27289421
- [Derived] Singh L, Garate B, Hoppe JM, Holmes EA. Qualitative analysis of hotspots and intrusive memories after viewing an aversive film highlights their sensory and spatial features. Sci Rep. 2022 Apr 29;12(1):7049. doi: 10.1038/s41598-022-10579-0. PMID 35487945